CLINICAL TRIAL: NCT02597543
Title: Stress Cardiac MRI Using Regadenoson for Evaluation of Nonspecific Allograft Dysfunction
Brief Title: Stress Cardiac MRI for Evaluation of Nonspecific Allograft Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul Kim (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Paul Kim, Cardiology Fellow, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1186278
Record Dates: First submitted 2015-10-30; First posted 2015-11-05 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-07

CONDITIONS: Heart Transplant; Acute Graft Rejection; Chronic Graft Rejection
Keywords: heart transplantation; cardiac MRI; graft rejection; nonspecific allograft dysfunction; allograft vasculopathy
MeSH Terms: interventions — regadenoson; Gadolinium; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonspecific allograft dysfunction (Experimental): Patients with nonspecific allograft dysfunction will undergo stress cardiac MRI with regadenoson in addition to performing late gadolinium enhancement and obtaining mean segmental T1 values of the heart.
  Interventions: Drug: Regadenoson; Drug: Gadolinium; Procedure: Cardiac MRI
- Normal graft function (Experimental): Patients with normal graft function will undergo stress cardiac MRI with regadenoson in addition to performing late gadolinium enhancement and obtaining mean segmental T1 values of the heart.
  Interventions: Drug: Regadenoson; Drug: Gadolinium; Procedure: Cardiac MRI

INTERVENTIONS:
Drug: Regadenoson — For use in stress myocardial perfusion imaging.
  Other Names: Lexiscan
Drug: Gadolinium — For use in both perfusion imaging and late gadolinium enhancement.
  Other Names: Magnevist
Procedure: Cardiac MRI — Cardiac MRI will be the imaging modality for perfusion imaging, late gadolinium enhancement and obtaining mean T1 segmental values of the heart.

SUMMARY:
The investigators will use cardiac MRI to measure the myocardial perfusion reserve and amount of myocardial edema and fibrosis in heart-transplant patients with nonspecific allograft dysfunction in contrast to those with normal graft function. The investigators hypothesize that patients with nonspecific allograft dysfunction will demonstrate decreased myocardial perfusion reserve, related to microvascular allograft vasculopathy, compared to those with normal graft function.

DETAILED DESCRIPTION:
Adult heart-transplant patients, excluding those with a GFR less than 30 mL/min/1.73m2, contraindications to MRI and allergies to either regadenoson or gadolinium contrast, will be enrolled over 10 months. Patients will be recruited from UC San Diego and San Diego Veterans Affairs. The investigators will specifically enroll patients with nonspecific allograft dysfunction and patients with normal graft function.

Brief protocol:

Cardiac MRI is performed. Cine images in standard views are obtained. T2 mapping sequences are performed on short axis images. For stress imaging, intravenous regadenoson is given as a 0.4 mg bolus followed by a 5 mL saline flush. After 30 seconds, short-axis images are acquired for 30 consecutive heartbeats with administration of gadolinium. Rest imaging is performed 30 minutes after stress imaging. Lastly, late gadolinium enhancement images are obtained in standard views. Images are analyzed offline by a blinded independent reader. Patients will be followed for one month after enrollment for MACE.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* At least three months status post heart transplantation.
* Heart-transplant patients with normal graft function (left ventricular ejection fraction equal to or greater than 55%) and no prior history of clinically significant acute rejection episodes that required modification of the immunosuppressive regimen or cardiac allograft vasculopathy.
* Heart-transplant patients with nonspecific allograft dysfunction (left ventricular ejection fraction equal to or less than 50% AND decrease from post-transplant baseline ejection fraction by an absolute difference of 10% or greater, no formal diagnosis of allograft vasculopathy by coronary angiogram or coronary vascular ultrasonography, and no history of prior acute rejection episodes known to have decreased left ventricular ejection fraction to or less than 50%).

Exclusion Criteria:

* Biopsy proven acute rejection episode in the past 3 months.
* Patients with symptoms or signs of acute myocardial ischemia or recent acute coronary syndrome in the past 3 months.
* Uncontrolled obstructive ventilatory disease including asthma and COPD.
* Second or third degree AV nodal block.
* Sinus node dysfunction.
* Contraindications to MRI including pacemakers or implantable cardioverter-defibrillators.
* Renal dysfunction with an estimated GFR less than 30 mL/min/1.73m2.
* Prior adverse reaction to either regadenoson or gadolinium contrast. Prior adverse reaction to adenosine will be assessed on a case-by-case basis.
* Any invasive procedure, including endomyocardial biopsy and left coronary angiogram, performed within one week.
* Systolic blood pressure greater than 180 or less than 85 mmHg.
* Diastolic blood pressure greater than 120 or less than 40 mmHg.
* Resting heart rate greater than 120 or less than 45 beats per minute.
* Severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Kim, MD, Principal Investigator — Stanford University
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Stehlik J, Edwards LB, Kucheryavaya AY, Benden C, Christie JD, Dobbels F, Kirk R, Rahmel AO, Hertz MI. The Registry of the International Society for Heart and Lung Transplantation: Twenty-eighth Adult Heart Transplant Report--2011. J Heart Lung Transplant. 2011 Oct;30(10):1078-94. doi: 10.1016/j.healun.2011.08.003. No abstract available. PMID 21962016
- [Background] Berry GJ, Angelini A, Burke MM, Bruneval P, Fishbein MC, Hammond E, Miller D, Neil D, Revelo MP, Rodriguez ER, Stewart S, Tan CD, Winters GL, Kobashigawa J, Mehra MR. The ISHLT working formulation for pathologic diagnosis of antibody-mediated rejection in heart transplantation: evolution and current status (2005-2011). J Heart Lung Transplant. 2011 Jun;30(6):601-11. doi: 10.1016/j.healun.2011.02.015. No abstract available. PMID 21555100
- [Background] Costanzo MR, Dipchand A, Starling R, Anderson A, Chan M, Desai S, Fedson S, Fisher P, Gonzales-Stawinski G, Martinelli L, McGiffin D, Smith J, Taylor D, Meiser B, Webber S, Baran D, Carboni M, Dengler T, Feldman D, Frigerio M, Kfoury A, Kim D, Kobashigawa J, Shullo M, Stehlik J, Teuteberg J, Uber P, Zuckermann A, Hunt S, Burch M, Bhat G, Canter C, Chinnock R, Crespo-Leiro M, Delgado R, Dobbels F, Grady K, Kao W, Lamour J, Parry G, Patel J, Pini D, Towbin J, Wolfel G, Delgado D, Eisen H, Goldberg L, Hosenpud J, Johnson M, Keogh A, Lewis C, O'Connell J, Rogers J, Ross H, Russell S, Vanhaecke J; International Society of Heart and Lung Transplantation Guidelines. The International Society of Heart and Lung Transplantation Guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2010 Aug;29(8):914-56. doi: 10.1016/j.healun.2010.05.034. No abstract available. PMID 20643330
- [Background] Uretsky BF, Murali S, Reddy PS, Rabin B, Lee A, Griffith BP, Hardesty RL, Trento A, Bahnson HT. Development of coronary artery disease in cardiac transplant patients receiving immunosuppressive therapy with cyclosporine and prednisone. Circulation. 1987 Oct;76(4):827-34. doi: 10.1161/01.cir.76.4.827. PMID 3308166
- [Background] Fang JC, Kinlay S, Beltrame J, Hikiti H, Wainstein M, Behrendt D, Suh J, Frei B, Mudge GH, Selwyn AP, Ganz P. Effect of vitamins C and E on progression of transplant-associated arteriosclerosis: a randomised trial. Lancet. 2002 Mar 30;359(9312):1108-13. doi: 10.1016/S0140-6736(02)08154-0. PMID 11943259
- [Background] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- [Background] Bhalodolia R, Cortese C, Graham M, Hauptman PJ. Fulminant acute cellular rejection with negative findings on endomyocardial biopsy. J Heart Lung Transplant. 2006 Aug;25(8):989-92. doi: 10.1016/j.healun.2006.04.002. Epub 2006 Jun 30. PMID 16890123
- [Background] Miller CA, Sarma J, Naish JH, Yonan N, Williams SG, Shaw SM, Clark D, Pearce K, Stout M, Potluri R, Borg A, Coutts G, Chowdhary S, McCann GP, Parker GJ, Ray SG, Schmitt M. Multiparametric cardiovascular magnetic resonance assessment of cardiac allograft vasculopathy. J Am Coll Cardiol. 2014 Mar 4;63(8):799-808. doi: 10.1016/j.jacc.2013.07.119. Epub 2013 Dec 18. PMID 24355800
- [Background] Marie PY, Angioi M, Carteaux JP, Escanye JM, Mattei S, Tzvetanov K, Claudon O, Hassan N, Danchin N, Karcher G, Bertrand A, Walker PM, Villemot JP. Detection and prediction of acute heart transplant rejection with the myocardial T2 determination provided by a black-blood magnetic resonance imaging sequence. J Am Coll Cardiol. 2001 Mar 1;37(3):825-31. doi: 10.1016/s0735-1097(00)01196-7. PMID 11693758
- [Background] Butler CR, Thompson R, Haykowsky M, Toma M, Paterson I. Cardiovascular magnetic resonance in the diagnosis of acute heart transplant rejection: a review. J Cardiovasc Magn Reson. 2009 Mar 12;11(1):7. doi: 10.1186/1532-429X-11-7. PMID 19284612
- [Background] Kubrich M, Petrakopoulou P, Kofler S, Nickel T, Kaczmarek I, Meiser BM, Reichart B, von Scheidt W, Weis M. Impact of coronary endothelial dysfunction on adverse long-term outcome after heart transplantation. Transplantation. 2008 Jun 15;85(11):1580-7. doi: 10.1097/TP.0b013e318170b4cd. PMID 18551063
- [Background] Solberg OG, Ragnarsson A, Kvarsnes A, Endresen K, Kongsgard E, Aakhus S, Gullestad L, Stavem K, Aaberge L. Reference interval for the index of coronary microvascular resistance. EuroIntervention. 2014 Jan 22;9(9):1069-75. doi: 10.4244/EIJV9I9A181. PMID 24457279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 3 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [48 to 70.5] | 66 [52 to 68.5] | 64 [48 to 70.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion Reserve
Description: Myocardial perfusion reserve calculates the increase in myocardial perfusion after stress in comparison to rest. Outcome measure time frame specifies when the myocardial perfusion reserve was obtained in relation to date of heart-transplant for each patient. This was a one time measurement made after heart-transplantation.
Time Frame: Range of 1 to 12 years after heart transplantation for subjects and an average of 4 years after heart-transplantation.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
arbitrary units | 1.52 (0.52) | 1.94 (0.37)

2. Secondary Outcome: Myocardial Ischemia/Infarction
Description: Myocardial ischemia or infarct occurring from time of enrollment (when cardiac MRI performed) over subsequent 10 month period.
Time Frame: 10 months after enrollment (when cardiac MRI was performed)
Measure: Count of Participants; unit: Participants
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

3. Secondary Outcome: Hospitalization for Cardiac Related Causes
Description: Hospitalization for cardiac related causes after enrollment. Time frame after enrollment (date of cardiac MRI) was 10 months
Time Frame: 10 months after enrollment (from date of cardiac MRI)
Measure: Count of Participants; unit: Participants
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

4. Secondary Outcome: Re-transplantation
Description: Re-transplantation of the heart after enrollment (date of cardiac MRI). Measured 10 months after enrollment.
Time Frame: 10 months after enrollment (from date of cardiac MRI)
Measure: Count of Participants; unit: Participants
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

5. Secondary Outcome: Late Gadolinium Enhancement
Description: Late gadolinium enhancement demonstrates myocardial scar by cardiac MRI. This is measured the day of the cardiac MRI scan and is a one time measurement. Time frame is measurement of late gadolinium enhancement from date of heart-transplantation.
Time Frame: Range of 1 to 12 years after heart transplantation for subjects and an average of 4 years after heart-transplantation.
Measure: Mean (Standard Deviation); unit: percentage of myocardium
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
percentage of myocardium | 5.7 (2.6) | 1.8 (0.8)

6. Secondary Outcome: Mean Segmental T1 Values of the Left Ventricle
Description: T1 values are obtained at the time of the cardiac MRI and indicate the amount of myocardial edema. This was a one time measurement. Outcome measure time frame indicates when T1 values of the left ventricle were obtained in relation to heart-transplantation.
Time Frame: Range of 1 to 12 years after heart transplantation for subjects and an average of 4 years after heart-transplantation.
Measure: Mean (Standard Deviation); unit: Percentage of myocardium
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
Number analyzed (Participants) | 6 | 8
Percentage of myocardium | 44.5 (6.3) | 38.1 (5.9)

ADVERSE EVENTS:
Arm/Group | Nonspecific Allograft Dysfunction | Normal Graft Function
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No